CLINICAL TRIAL: NCT03630913
Title: Sentinel Lymph Node After Neoadjuvant Chemotherapy in Breast Carcinoma
Acronym: GANEA3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2018-03
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Invasive Breast Cancer; Axillary Metastases
Keywords: Neoadjuvant chemotherapy; Sentinel lymph node; Axillary lymphadenectomy; Tagged axillary metastatic node

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tagged axillary metastatic node (Experimental): Patients undergo axillary sonography assessment routinely performed to seek suspicious nodes. A cytological examination (biopsy is optional) of the suspicious node is performed.
  The involved node is then tagged with a metal clip under sonography. Then, patients receive NAC before surgery. Breast surgery (conservative or radical) and axillary surgery are performed during the same procedure, 4 to 6 weeks after completion of NAC.
  Interventions: Procedure: Tagged axillary metastatic node

INTERVENTIONS:
Procedure: Tagged axillary metastatic node — First, initially metastatic lymph node is tagged with a metal clip under sonography. Then, patients receive NAC before surgery.
  Breast surgery (conservative or radical) and axillary surgery are performed during the same procedure, 4 to 6 weeks after completion of NAC.
  SLN isotope detection is performed with or without blue dye. All patients undergo the resection of the tagged axillary node, SLN biopsy and a complementary axillary lymphadenectomy.

SUMMARY:
Sentinel lymph node dissection (SLND) after NAC, aimed to reduce the rate of unnecessary axillary lymphadenectomy, is not a standard of care in case of patient with previously involved node before NAC because of a too high false negative rate (FNR).

Clinical consequences of FNR of SLND after NAC are currently unknown. Consequently, contrary to adjuvant setting, a risk of SLND false negative case after NAC is not acceptable.

GANEA3 aims to evaluate the results of an innovative multiparametric strategy combining (1) an identification before chemotherapy of a lymph node involvement using a metal clip and then its analysis after treatment, (2) the analysis of sentinel lymph node (SLN) after NAC, and (3) analysis of biological parameters of breast tumor before and after NAC, to predict axillary status after NAC. This will identify patients with initial lymph node involvement who could benefit from SLN after NAC without additional axillary dissection with a very low FNR (≤1%).

The most "pathological" metastatic lymph node will be identified with a metal clip under ultrasound. They will then receive a NAC before breast and axillary surgery. An assessment of the NAC response at the breast and axillary will be performed by imagery. Then, all patients undergo the resection of the tagged axillary node with the metal clip, SLN detection and biopsy and a complementary axillary lymphadenectomy.

DETAILED DESCRIPTION:
GANEA3 is a prospective multicenter diagnostic study assessing the benefit of targeting initial involved node in complement to SLND and breast tumor characteristics to predict axillary status after NAC.

The diagnostic performances of this strategy will be primarily assessed by the decrease of the FNR with the combined strategy compared to SLND alone.

The primary objective is to evaluate the interest of identifying, before NAC, the initial involved lymph node to improve the prediction of axillary status after NAC.

The main secondary objectives are :

* To assess the feasibility, at the time of the surgery, of the identification and resection of the initially involved lymph node, tagged with the metal clip before NAC ;
* To evaluate the complications related to the setting up of the metal clip for the identification of a lymph node metastatic ;
* To evaluate the interest and impact of immunohistochemical analysis of tagged lymph node and SLN ;

Patients treated for a large early breast cancer (BC) needing NAC undergo axillary sonography assessment routinely performed to seek suspicious nodes. When several suspicious nodes are found only the worst is chosen. A fine needle aspiration is performed to allow cytological examination (biopsy is optional) of the suspicious node. In case of proven axillary involvement, the patient is informed about GANEA 3 study in order to be included.

At this step the patient must accept the study and sign the consent form. The involved node is then tagged (with a metal clip) under sonography. In case of multiple suspicious nodes, the radiologist must choose the worst node in order to tag only one involved node.

Then, then patients will perform their chemotherapy. The choice of NAC regimen is let at the discretion of each participating team.

After NAC, breast tumor size and axillary assessment are performed.

Breast and axillary surgery are performed during the same procedure, 4 to 6 weeks after completion of NAC. Breast surgery can be conservative or radical.

All patients undergo the resection of the tagged axillary node, SLN biopsy and a complementary axillary lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Initial diagnosis of operable invasive breast carcinoma
3. Histologically proven axillary metastasis (cytology or biopsy) before NAC
4. Patient included in a therapeutic approach of neoadjuvant chemotherapy
5. Procedure for the detection of sentinel lymph node by isotopic method +/- colorimetric
6. Information of the patient and obtaining written consent, signed by the patient and the investigator
7. Affiliated patient or beneficiary of the social security

Exclusion Criteria:

1. pT4d (inflammatory breast cancer)
2. Metastatic breast cancer
3. Any prior chemotherapy for contralateral breast cancer
4. Local relapse of breast cancer
5. Axillary metastasis not histologically proven before NAC
6. Allergy known to the 2 detection products (Blue and radioactive tracer)
7. Pregnant or lactating woman
8. Neo Adjuvant chemotherapy contraindicated
9. Patient protected or under guardianship or unable to give consent
10. Impossibility of submitting to the medical examination for geographical, social or psychological

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
False negative rate | 30 days after surgery
  number of cases of false prediction of absence of lymph node involvement to the total number of cases with metastatic lymph node. The rate of FN will be calculated for the involved lymph node tagged with the metal clip, the sentinel node, and the both

SECONDARY OUTCOMES:
Identification rate of involved lymph node tagged | 30 days after surgery
  number of cases where the tagged lymph node with a metal clip node is identified during axillary surgery and analyzed in pathology on the total number of procedures
Resection rate of involved lymph node tagged | 30 days after surgery
  number of cases where the tagged lymph node is resected during axillary surgery and analyzed in pathology on the total number of procedures
Complication rate | 30 days after surgery
  number of complications related to the axillary lymph node tagging procedure on the total number of procedures

CONTACTS AND LOCATIONS:
Overall Officials: JEAN-MARC CLASSE, MD, Study Director — ICO NANTES
Locations (18):
- France (18):
  - ICO - Site ANGERS, Angers
  - Institut Bergonié, Bordeaux
  - CHU Brest, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francoise Leclerc, Dijon
  - Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Montpellier, Montpellier
  - APHP - Pitié Salpétrière, Paris
  - Hôpital St JOSEPH, Paris
  - Anne-Sophie Georges BATS, Paris
  - Centre Jean Godinot, Reims
  - CURIE, Saint-Cloud
  - CHP St GREGOIRE, Saint-Grégoire
  - Céline RENAUDEAU, Saint-Herblain
  - IUCT-O, Toulouse
  - Institut de Cancérlogie de Lorraine, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Ditsch N, Rubio IT, Gasparri ML, de Boniface J, Kuehn T. Breast and axillary surgery in malignant breast disease: a review focused on literature of 2018 and 2019. Curr Opin Obstet Gynecol. 2020 Feb;32(1):91-99. doi: 10.1097/GCO.0000000000000593. PMID 31833973